CLINICAL TRIAL: NCT00757965
Title: A Population Based Study of Genetic Predisposition and Gene-Environment Interactions in Colorectal Cancer in East Anglia
Brief Title: Study of Genes and the Environment in Patients With Colorectal Cancer in the East Anglia Region of the United Kingdom
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cancer Research UK (Other)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: CDR0000598882; MREC-SEARCH-COLORECTAL; MREC-07/MRE05/17
Record Dates: First submitted 2008-09-22; First posted 2008-09-23 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2008-09

CONDITIONS: Colorectal Cancer
Keywords: colon cancer; rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Amplified Fragment Length Polymorphism Analysis

INTERVENTIONS:
Genetic: polymorphism analysis
Other: laboratory biomarker analysis
Other: questionnaire administration

SUMMARY:
RATIONALE: Studying samples of blood from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This study is looking at genetic susceptibility for cancer and interactions between genes and the environment in patients with colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To obtain epidemiological information and biological material on a population based series of colorectal cancer cases.
* To define the proportion of colorectal cancer incidence attributable to mutations in known predisposing genes such as MLH1 and MSH2.
* To establish whether mutations at other loci may predispose to colorectal cancer, by comparing the frequency of alteration candidate genes in colorectal cancer patients with the corresponding frequency in cancer-free controls identified through the European Prospective Investigation of Cancer (EPIC) study.

OUTLINE: This is a multicenter study.

Patients complete an epidemiological questionnaire. The questionnaire also requests identifying information about the patient's first-degree relatives.

Blood samples are collected from patients. DNA is extracted from these blood samples, from samples collected from cancer-free control participants in MREC-SEARCH-CONTROL, and from additional controls through the European Prospective Investigation of Cancer (EPIC) study (a population-based study of diet and health based in Norfolk, East Anglia). DNA samples are analyzed for polymorphisms of low penetrance cancer susceptibility genes.

In addition to the colorectal cancer patients recruited for this study, patients with breast, ovarian, prostate, colorectal, bladder, kidney, pancreatic, brain, and esophageal cancer, malignant melanoma, and lymphoma cancer are recruited for the following related clinical trials: MREC-SEARCH-BREAST, MREC-SEARCH-OVARIAN, MREC-SEARCH-PROSTATE, MREC-SEARCH-ENDOMETRIAL, and MREC-SEARCH-CANCER.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of colorectal cancer within the past 5 years
* Identified in the East Anglia region of the United Kingdom

PATIENT CHARACTERISTICS:

* Identified by the patient's general practitioner as fit to contact for this study
* No serious mental illness or retardation

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2008-02

PRIMARY OUTCOMES:
Acquisition of epidemiological information and biological material
Proportion of colorectal cancer incidence attributable to mutations in known predisposing genes (e.g., MLH1 and MSH2)
Exploration of mutations at other loci that may predispose to endometrial cancer

CONTACTS AND LOCATIONS:
Overall Officials: Paul Pharoah, MD, Study Chair — Cancer Research UK
Locations (1):
- University of Cambridge Cancer Research UK, Cambridge, England, United Kingdom